CLINICAL TRIAL: NCT00358982
Title: A Phase II Study of MGCD0103 (MG-0103) in Patients With Relapsed or Refractory Hodgkin's Lymphoma
Brief Title: Study of MGCD0103 (MG-0103) in Patients With Relapsed or Refractory Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0103-010
Record Dates: First submitted 2006-07-31; First posted 2006-08-01 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-06

CONDITIONS: Hodgkin's Lymphoma
Keywords: Relapsed or Refractory Hodgkin's Lymphoma; Phase II
MeSH Terms: conditions — Hodgkin Disease; Recurrence | interventions — mocetinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: MGCD0103

INTERVENTIONS:
Drug: MGCD0103 — MGCD0103 administered orally three times per wek

SUMMARY:
MGCD0103 is an experimental drug that belongs to a class of drugs known as the histone deacetylase inhibitors, which may restore normal control in cancer cells by affecting the genes and proteins that are being made. Laboratory tests show that this new investigational anti-cancer drug can slow down the growth of human cancer cells in mice; two clinical research studies are currently being performed in humans with cancer and a similar study is being performed in patients with the same disease.

The purpose of this study is to find out what effect the experimental drug MGCD0103 has on patients with relapsed and refractory Hodgkin's lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic confirmation of relapsed or refractory classical Hodgkin's lymphoma.
* The patient has at least one site of measurable disease (≥ 2.0 cm) as measured by conventional techniques such as CT or MRI.
* Prior treatment: there is no limit to number of prior therapies. Patients who had prior allogeneic stem cell transplants and do not have evidence of graft versus host disease and are not receiving immunosuppressive agents are eligible if they meet all other inclusion criteria.
* ECOG performance status of 0 or 1.
* Aged 18 years or older (no safety data yet for ages < 18).
* Laboratory requirements (must be done within 7 days prior to study initiation).

Exclusion Criteria:

* Patients with another active cancer (excluding basal cell carcinoma or cervical intraepithelial neoplasia [CIN/cervical in situ] or melanoma in situ). Prior history of cancer is allowed, as long as there is no active disease.
* Pregnant or lactating women. Women of child-bearing potential (WOCBP) must have a negative serum pregnancy test documented within 7 days prior to start of study drug.
* WOCBP and men whose partners are WOCBP must use an acceptable method of contraception while enrolled in this study, and for a period of 3 months following study drug treatment.
* Patients with uncontrolled intercurrent illness, active or uncontrolled infections, or a fever > 38.5°C (not due to tumor fever) on the day of scheduled dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2006-08; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Success rate | 1 year (anticipated)

SECONDARY OUTCOMES:
Progression-free survival | 1 year (anticipated)
Duration of objective response | 1 year (anticipated)
Safety profile | 1 year (anticipated)
Pharmacodynamics (biomarkers) | 1 year (anticipated)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Reid, MSc, MBA, Study Director — MethylGene Inc.
Locations (5):
- United States (3):
  - Rush University Medical Center, Chicago, Illinois
  - Nebraska Medical Center, Omaha, Nebraska
  - MD Anderson Cancer Center, Houston, Texas
- Canada (2):
  - Princess Margaret Hospital, Toronto, Ontario
  - Royal Victoria Hospital, Montreal, Quebec

REFERENCES:
- [Derived] Younes A, Oki Y, Bociek RG, Kuruvilla J, Fanale M, Neelapu S, Copeland A, Buglio D, Galal A, Besterman J, Li Z, Drouin M, Patterson T, Ward MR, Paulus JK, Ji Y, Medeiros LJ, Martell RE. Mocetinostat for relapsed classical Hodgkin's lymphoma: an open-label, single-arm, phase 2 trial. Lancet Oncol. 2011 Dec;12(13):1222-8. doi: 10.1016/S1470-2045(11)70265-0. Epub 2011 Oct 25. PMID 22033282